CLINICAL TRIAL: NCT00669318
Title: Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL) With Pentostatin, Alemtuzumab, and Low Dose Rituximab: A Phase II Clinical Trial
Brief Title: Pentostatin, Alemtuzumab, and Rituximab in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS0881; LS0881 (Other: Mayo Clinic Cancer Center); 08-000673 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-04-29; First posted 2008-04-30 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; Pentostatin; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Pentostatin, Alemtuzumab, Rituximab) (Experimental): Course 1: Patients receive:
  * 2 mg/m^2 pentostatin IV on days 8 and 22;
  * 3 mg alemtuzumab subcutaneously (SC) on day 3;
  * 10 mg alemtuzumab SC on day 4;
  * 30 mg alemtuzumab SC on days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  * 20 mg/m^2 rituximab IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  * 6 mg Sargramostim (GM-CSF) SC on days 10-14. Patients then proceed to course 2.
  Courses 2 and 3: Patients receive:
  * 2 mg/m^2 pentostatin IV on days 1 and 15;
  * 30 mg alemtuzumab SC on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26;
  * 20 mg/m^2 rituximab IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26;
  * 6 mg GM-CSF SC on days 3-7. After completion of course 2, patients with a complete response proceed to observation. Patients with a partial response or stable disease receive another course of therapy (course 3).
  Interventions: Biological: alemtuzumab; Biological: rituximab; Drug: pentostatin; Drug: sargramostim

INTERVENTIONS:
Biological: alemtuzumab
Biological: rituximab
Drug: pentostatin
Drug: sargramostim
  Other Names: GM-CSF

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pentostatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as alemtuzumab and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving pentostatin together with alemtuzumab and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving pentostatin together with alemtuzumab and rituximab works in treating patients with relapsed or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the rate of complete and overall response in patients with relapsed or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma treated with pentostatin, alemtuzumab, and low-dose rituximab.
* To monitor and assess toxicity of this treatment regimen.

Secondary

* To determine the overall and progression-free survival, duration of response, and time to next treatment.
* To assess the correlation between individual prognostic markers (17p-, 11q-, unmutated VH gene, VH3-21, ZAP-70+, CD38+, CD49d, and β2 microglobulin, miRNA profiles, angiogenesis status, and karyotypes of CpG stimulated cells) and clinical outcome.

OUTLINE: This is a multicenter study.

* Course 1: Patients receive pentostatin IV on days 8 and 22; alemtuzumab subcutaneously (SC) on days 3-5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33; rituximab IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33; and sargramostim (GM-CSF) SC on days 10-14 and 24-28. Patients then proceed to course 2.
* Courses 2 and 3: Patients receive pentostatin IV on days 1 and 15; alemtuzumab SC and rituximab IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26; and GM-CSF SC on days 3-7 and 17-21. After completion of course 2, patients with a complete response proceed to observation. Patients with a partial response or stable disease receive another course of therapy (course 3).

Treatment continues in the absence of disease progression or unacceptable toxicity.

Blood is collected on days 1, 3, 8, and 10 of course 1 for monoclonal antibody studies. Samples are analyzed for serum concentration of alemtuzumab and rituximab by ELISA and PCR; CH50 assay; complement activation and cytokine levels by ELISA; NK cell activation; and NK cell phenotype by immunofluorescent staining and flow cytometry.

After completion of study treatment, patients are followed up monthly for 6 months, every 3 months for 6 months, and then every 6-12 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) meeting the following criteria:

  * Minimum threshold peripheral blood lymphocyte count of 5 x 10^9/L (CLL variant) OR adenopathy > 1 cm or palpable splenomegaly (SLL variant)
  * Immunophenotypic demonstrations of a population of B lymphocytes (as defined by CD19+) that are monoclonal (by light chain exclusion) AND have ≥ 3 of the following characteristics:

    * CD5+
    * CD23+
    * Dim surface light chain expression
    * Dim surface CD20 expression
    * FISH analysis is negative for IGH/CCND1 and/or immunostaining is negative for cyclin D1 expression
* Must have progressive disease as indicated by any of the following characteristics (based on standard criteria for treatment):

  * Symptomatic CLL characterized by any of the following:

    * Weight loss > 10% within the past 6 months
    * Extreme fatigue
    * Fevers > 38.5° C (not due to infection)
    * Drenching night sweats without evidence of infection
  * Evidence of progressive bone marrow failure with hemoglobin < 11 g/dL or platelet count < 100 x 10^9/L
  * Massive and progressive splenomegaly (> 6 cm below left costal margin)
  * Massive (> 10 cm) or rapidly progressive lymphadenopathy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Creatinine ≤ 2 times upper limit of normal (ULN)
* Total bilirubin ≤ 3.0 times ULN OR direct bilirubin ≤ 1.5 times ULN
* AST ≤ 3.0 times ULN (unless due to hemolysis or CLL)
* Willing to provide mandatory blood samples for research studies
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 12 months after completion of study treatment
* No other active primary malignancy that requires treatment or limits survival to ≤ 2 years
* No active autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past month
* No uncontrolled infection
* No HIV infection or AIDS
* No active hepatitis B infection (i.e., HBsAg or HBeAg positivity) or hepatitis C infection by serology
* No other comorbid condition

PRIOR CONCURRENT THERAPY:

* No more than 3 prior treatment regimens for CLL that included purine analogue drugs (e.g., fludarabine, pentostatin, or cladribine) OR previously untreated CLL in patients with high-risk disease due to 17p13 deletion on FISH analysis
* More than 4 weeks since prior major surgery
* More than 2 months since prior alemtuzumab
* Prior corticosteroids allowed
* No concurrent continuous systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-07; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clive S. Zent, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Zent CS, Taylor RP, Lindorfer MA, Beum PV, LaPlant B, Wu W, Call TG, Bowen DA, Conte MJ, Frederick LA, Link BK, Blackwell SE, Veeramani S, Baig NA, Viswanatha DS, Weiner GJ, Witzig TE. Chemoimmunotherapy for relapsed/refractory and progressive 17p13-deleted chronic lymphocytic leukemia (CLL) combining pentostatin, alemtuzumab, and low-dose rituximab is effective and tolerable and limits loss of CD20 expression by circulating CLL cells. Am J Hematol. 2014 Jul;89(7):757-65. doi: 10.1002/ajh.23737. Epub 2014 Apr 26. PMID 24723493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-one patients were enrolled from July 2008 to February 2013 and 39 were evaluable. Two patients did not start treatment. One patient was found to have concomitant Hodgkin lymphoma and the other a serious systemic infection during pre-treatment evaluation. The characteristics of the 39 evaluable patients are summarized
Period: Overall Study
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Started | 41
Completed | 39
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: A Complete Response (CR) requires the disappearance of all nodes, a non-palpable liver and spleen, no constitutional symptoms, absolute neutrophil counts >1500/uL, platelets >100000/uL, Hemoglobin >11.0 g/dL, and lymphocytes <4000/uL. In addition, a bone marrow biopsy with evidence of <30% lymphocytes and no nodules.
  Here we report the rate of complete response as the number of patients attaining a CR status divided by the total number of evaluable patients. The 95% CI is estimated using the binomial distribution.
Time Frame: Up to 3 cycles of treatment and 2 cycles of observation (up to 5 months total)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
percentage of participants | 10 [2.9 to 24.2]

2. Secondary Outcome: Overall Response Rate (Complete and Partial Response)
Description: A Complete Response (CR) requires the disappearance of all nodes, a non-palpable liver and spleen, no constitutional symptoms, absolute neutrophil counts >1500/uL, platelets >100000/uL, Hemoglobin >11.0 g/dL, and lymphocytes <4000/uL. A bone marrow biopsy with evidence of <30% lymphocytes and no nodules.
  Patients who fulfill all criteria for a CR but have a persistent anemia, thrombocytopenia, or neutropenia related to drug toxicity will be classified as CR with incomplete marrow recovery (CRi).
  A Partial Response (PR) requires a 50% reduction in nodes and liver/spleen measurements and at least two of the following: absolute neutrophil counts >1500/uL, platelets >100000/uL, Hemoglobin >11.0 g/dL, or a >50% reduction in lymphocytes.
  Here we report the rate of overall response as the number of patients attaining a CR, PR, or CRi status divided by the total number of evaluable patients. The 95% CI is estimated using the binomial distribution.
Time Frame: Up to 3 cycles of treatment and 2 cycles of observation (up to 5 months total)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
percentage of patients | 56 [40 to 72]

3. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Follow-up status and retreatment information will be collected up to 5 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
months | 34.1 [13.6 to NA] — A sufficient number of events has not occurred to accurately estimate the 95% confidence interval.

4. Secondary Outcome: Progression-free Survival
Description: The progression-free survival (PFS) time is defined as the time from registration to progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Follow-up status and retreatment information will be collected up to 5 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
months | 7.2 [5.3 to 18.3]

5. Secondary Outcome: Time to Retreatment
Description: Time to subsequent therapy is defined to be the time from the registration to the date subsequent therapy is initiated. The distribution of time to subsequent therapy will be estimated using the method of Kaplan-Meier
Time Frame: Follow-up status and retreatment information will be collected up to 5 years from registration
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Number analyzed (Participants) | 39
months | 9.1 [5.7 to 27]

ADVERSE EVENTS:
Groups:
- Treatment (Pentostatin, Alemtuzumab, Rituximab): sargramostim
Arm/Group | Treatment (Pentostatin, Alemtuzumab, Rituximab)
Serious Adverse Events (participants affected / at risk) | 4/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pentostatin, Alemtuzumab, Rituximab) (N=39)
Pneumonia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pentostatin, Alemtuzumab, Rituximab) (N=39)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 22 (44)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Chills (General disorders) | 9 (12)
Edema limbs (General disorders) | 1 (2)
Fatigue (General disorders) | 10 (14)
Fever (General disorders) | 24 (40)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 4 (6)
Mucosal infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 11 (14)
Pneumonia (Infections and infestations) | 3 (7)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (4)
Skin infection (Infections and infestations) | 5 (6)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 30 (89)
Lymphocyte count decreased (Investigations) | 10 (31)
Neutrophil count decreased (Investigations) | 27 (58)
Platelet count decreased (Investigations) | 16 (34)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Seizure (Nervous system disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 17 (34)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes